CLINICAL TRIAL: NCT04271488
Title: An Open-label Parallel-Group Study to Evaluate Pharmacokinetics of E7090 and Its Metabolite in Subjects With Mild and Moderate Hepatic Impairment Compared to Healthy Subjects
Brief Title: Study to Evaluate the Pharmacokinetics (PK) of E7090 (Herein Referred to as Tasurgratinib) and Its Metabolite in Participants With Mild and Moderate Hepatic Impairment Compared to Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7090-J081-001
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; E7090; Tasurgratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A: Mild Hepatic Impairment (Child Pugh Class A) (Experimental): Participants with mild hepatic impairment will receive a single 35 milligram (mg) tablet of tasurgratinib in the morning with 150 milliliters (mL) of water following an overnight fast of at least 10 hours.
  Interventions: Drug: Tasurgratinib
- Cohort B: Moderate Hepatic Impairment (Child Pugh Class B) (Experimental): Participants with moderate hepatic impairment will receive 10 mg dose of tasurgratinib as capsule (2 capsules each of 5 mg) in the morning with 150 mL of water following an overnight fast of at least 10 hours.
  Interventions: Drug: Tasurgratinib
- Cohort C: Healthy Participants (Control) (Experimental): Healthy participants matched to participants with hepatic impairment in Cohorts A and B (matched with regards to age, race, gender and body weight) will receive a single 35 mg tablet of tasurgratinib in the morning with 150 mL of water following an overnight fast of at least 10 hours.
  Interventions: Drug: Tasurgratinib

INTERVENTIONS:
Drug: Tasurgratinib — Tasurgratinib oral tablet.
  Arms: Cohort A: Mild Hepatic Impairment (Child Pugh Class A); Cohort C: Healthy Participants (Control)
Drug: Tasurgratinib — Tasurgratinib oral capsule.
  Arms: Cohort B: Moderate Hepatic Impairment (Child Pugh Class B)

SUMMARY:
The primary purpose of the study is to evaluate the effects of mild and moderate hepatic impairment on PK of tasurgratinib after a single dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) between 18 to 40 kilogram per square meter (kg/m^2).
2. For Cohorts A and B: stable hepatic impairment conforming to Child-Pugh classification A and B.
3. For Cohort C: healthy participants matched to participants with hepatic impairment with regard to age (+/-10 years), body weight (+/-20 percent [%]), race and gender, and as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram (ECG), and clinical laboratory determinations.

Exclusion Criteria:

Key Exclusion for all Participants:

1. Following ocular disorders

   1. Current evidence of Grade 2 or higher corneal disorder
   2. Current evidence of active macular disorder (example, Age-related macular degeneration, central serous chorioretinal disease)
2. Known to be human immunodeficiency virus (HIV) positive at Screening.
3. A prolonged QT/QTc interval ([QT interval using Fridericia's formula] QTcF greater than (>) 480 millisecond [ms]) demonstrated on ECG.

Additional Exclusion Criteria for Hepatically Impaired Participants (Cohorts A and B)

In addition to the Exclusion Criteria above for all participants, other standard exclusion criteria for participants with hepatic impairment will be used. These include:

1. Any significant acute medical illness (such as new conditions or exacerbation of pre-existing conditions) within 8 weeks of dosing.
2. Presence of severe ascites, edema, or uncontrolled hepatic encephalopathy
3. The participant's standard therapy/concomitant medication for diseases related to hepatic disease has not remained stable/unchanged for at least two weeks before dosing of study drug.

Additional Exclusion Criteria for Healthy participants (Cohort C)

In addition to the Exclusion Criteria for all participants, other standard exclusion criteria for healthy participants in Phase 1 studies will be used. These include:

1. Syphilis as demonstrated by positive serology at Screening.
2. Any abnormal finding based on physical examination, assessment of vital signs, ECG, or laboratory test results that requires treatment or clinical follow up based on investigators opinion.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration of Tasurgratinib | Day 1: 0-144 hours postdose
AUC(0-t): Area Under the Plasma Concentration versus Time Curve from Time 0 to Time of Last Quantifiable Concentration of Tasurgratinib | Day 1: 0-144 hours postdose
AUC(0-inf): Area Under the Plasma Concentration versus Time Curve from Time 0 to Infinity of Tasurgratinib | Day 1: 0-144 hours postdose

SECONDARY OUTCOMES:
Tmax: Time to Reach Maximum Plasma Concentration of Tasurgratinib and its Metabolite | Day 1: 0-144 hours postdose
AUC(0-72Hours): Area Under the Plasma Concentration versus Time Curve from Time 0 to 72 Hours of Tasurgratinib and its Metabolite | Day 1: 0-144 hours postdose
T1/2: Terminal Phase Plasma Half-life of Tasurgratinib and its Metabolite | Day 1: 0-144 hours postdose
CL/F: Apparent Total Body Clearance of Tasurgratinib | Day 1: 0-144 hours postdose
Vz/F : Apparent Volume of Distribution at Terminal Phase of Tasurgratinib | Day 1: 0-144 hours postdose
AUC Metabolite Ratio: Ratio of AUC(0-inf) of M2 to AUC(0-inf) of Tasurgratinib, Corrected for Molecular Weights | Day 1: 0-144 hours postdose
fu: Plasma Protein Unbound Fraction of Tasurgratiniband its Metabolite | Day 1: 0-144 hours postdose
AUCu: AUC(0-inf) Values Adjusted by Unbound Fraction in Plasma of Tasurgratinib | Day 1: 0-144 hours postdose
CLu/F: Apparent Clearance Relative to the Unbound Plasma Concentration of Based on AUCu of Tasurgratinib | Day 1: 0-144 hours postdose

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Eisai Trial Site #6, Hakata, Fukuoka
  - Eisai Trial Site #4, Kurume, Fukuoka
  - Eisai Trial Site #2, Yuhu, Oita Prefecture
  - Eisai Trial Site #3, Bukyo-ku, Tokyo
  - Eisai Trial Site #1, Mintato-ku, Tokyo
  - Eisai Trial Site #8, Shinjuku-ku, Tokyo
  - Eisai Trial Site #5, Kofu, Yamanashi
  - Eisai Trial Site #7, Kyoto

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.